CLINICAL TRIAL: NCT00294554
Title: Double-Blind Placebo-Controlled Trial of Memantine for Treatment of Cognitive Impairment in Patients With Parkinson's Disease and Dementia
Brief Title: Memantine for Treatment of Cognitive Impairment in Patients With Parkinson's Disease and Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-08-20-03
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Parkinson's Disease; Cognitive Impairment; Dementia
Keywords: Parkinson's Disease; Cognitive Impairment; Dementia; Memory
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Dementia | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Memantine (Active Comparator): Memantine tablets, formulated in appearance to match the placebo comparator, were initiated at 5 mg daily and advanced by 5mg /week to 20 mg/week by week 4 with dosing at 10 mg bid over the remaining 20 weeks of the trial. Over the 6 month duration of the trial, dosage could be titrated downward in increments of 5 mg to a minimum dose of 5mg/day in the event of intolerance.
  Interventions: Drug: Memantine
- Placebo Oral Tablet (Placebo Comparator): Placebo tablets were formulated to match active 5mg memantine tablets. Dosing same as the active comparator with initiation at 5 mg daily and advancing by 5mg /week to 20 mg/week by week 4 with dosing at 10 mg bid over the remaining 20 weeks of the trial. Over the 6 month duration of the trial, dosage could be titrated downward in increments of 5 mg to a minimum dose of 5mg/day in the event of intolerance.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Memantine — Active memantine and placebo, taken by mouth, will be titrated from 5mg a day to 20mg a day over 4 weeks. The subject will remain on 20mg (10mg twice a day) through week 24 unless unable to tolerate. The dose will be decreased as needed.
  Other Names: Namenda
  Arms: Active Memantine
Drug: Placebo Oral Tablet — Placebo, taken by mouth, will be titrated from 5mg a day to 20mg a day over 4 weeks. The subject will remain on 20mg (10mg twice a day) through week 24 unless unable to tolerate. The dose will be decreased as needed.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this research is to evaluate the usefulness of memantine, compared to placebo (sugar pill), for the treatment of cognitive impairment in patients with idiopathic Parkinson's disease (PD) and dementia. Memantine is used as a safe and effective treatment for patients with Alzheimer's disease. Cognitive impairment includes concentration and memory difficulties. We will look at how well this medication helps your cognitive impairment, how well you tolerate this medication (including its effects on your motor symptoms of PD) your activities of daily living, your emotions, and any medical conditions you might have. We will interview a person you choose as your "informant".

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, parallel, double-blind 24-week prospective study of memantine at the dosage range 5-20 mg/day in 20 outpatients with idiopathic PD and dementia secondary to PD. Using the dosage escalation regimen approved for Alzheimer disease, subjects will start memantine or comparable placebo at 5 mg daily and advance 5 mg/week to 20 mg /day by week 4, with dosing at 10 mg bid. Subjects will undergo 7 clinical visits over the 6-month trial (Screen, Baseline/Week 0, and Weeks 4, 8, 14, 20, and 24). The dosage can be titrated downward in increments of 5 mg to a minimum dose of 5 mg/day in the event memantine is not tolerated at the scheduled dosages. This broad dose range is being used because 1)a favorable cognitive response may be evident at lower doses of memantine than recommended for AD and 2)adverse effects could emerge when typical AD dosing recommendations are used, as has been observed when treating PD patients with cholinesterase inhibitors. Subjects will remain on a stable dose of memantine/placebo after Week 8, unless precluded by adverse events. Ten subjects will be assigned to each treatment group. Randomization will be stratified according to whether subjects are taking a concomitant cholinesterase inhibitor. This will enable secondary group comparisons of treatment groups. Results from this initial small study will be used to evaluate the appropriateness of devising a larger-scale multi-site study of memantine for treatment of dementia in PD.

The proposed assessment schedule was designed to represent use of memantine in general clinical practice and to minimize the burdens to caregivers and patients, who have impaired mobility as well as cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD, as defined by UK Brain Bank Criteria.
2. Age onset of PD > 35 years old
3. Adult men and women, current age > 50 years
4. English speaking
5. Any race or ethnic background.
6. Hoehn and Yahr Stage I-V, provided able to participate verbally in clinical assessments and travel to clinic.
7. Diagnosis of dementia secondary to PD, as defined by DSM-IV-TR.
8. Stable medical health
9. Taking stable doses for 2 months of non-excluded medications.
10. Outpatient status (may be residing in a long-term care facility).
11. Able to attend all study visits with an informed caregiver/partner who is willing to provide information on the patient's clinical status and response to treatment.
12. Presence of an informed caregiver willing to take part in weekly phone call follow-up calls for the duration of study enrollment.
13. Provision of informed consent by patient and caregiver and/or legal guardian.
14. On stable antiparkinsonian therapy for 2 months.
15. If history of major depression or anxiety disorder, must have stable symptoms and be on stable therapy for 2 months.
16. If taking antipsychotic medication, must be on stable therapy for 2 months.
17. If taking nonsteroidal anti-inflammatory medication, selegiline, or estrogen, must be on a stable dose for 30 days before study entry.
18. If taking cholinesterase inhibitors, must be on for at least 6 months and a stable dose for 2 months before randomization.

Exclusion Criteria:

1. History or evidence of neurodegenerative disorder other than PD.
2. Meets clinical criteria for Dementia with Lewy Bodies.
3. History or current evidence of epilepsy.
4. Participation in another investigational drug trial within 2 months of screening.
5. Treatment with memantine within 60 days of screening.
6. Current symptomatic Major Depressive Disorder, as based on Hamilton Depression Rating Scale Score > 17.
7. Current clinically significant hepatic, kidney disease, gastrointestinal, endocrine, or cardiovascular disease, including evidence of second or third degree heart block. [Note, patients with controlled hypertension (supine diastolic BP<95 mm Hg), complete or partial right bundle branch block, pacemakers, or deep brain stimulators may be included.].

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marsh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women with idiopathic Parkinson's disease (PD) and dementia due to PD recruited from outpatient clinics at Johns Hopkins and outreach to the Baltimore-Washington community through the Johns Hopkins Morris K. Udall Parkinson's Disease Research Center. Recruitment period was 2006 to 2008.
Pre-assignment Details: Enrolled participants were excluded if screening assessment showed MMSE>10 and Clinical Dementia Rating (CDR) scale score >1, or diagnostic criteria for dementia with Lewy bodies or DSM-IV-TR substance abuse/dependence or major depressive episode, Hamilton Depression Rating Scale score>17, or severe cardiac, vascular or renal disease.
Period: Overall Study
Arm/Group | Active Memantine | Placebo Oral Tablet
Started | 10 | 10
Completed | 10 | 8 (1 S withdrew @ 20 wks for lack perceived benefit 1 S withdrawn @ 13 wks b/o extreme agitation)
Not Completed | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Memantine | Placebo Oral Tablet | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.3) | 71.9 (7.5) | 71.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Education [Mean (Standard Deviation); unit: years] | 17.2 (4.5) | 16.9 (3.0) | 17.1 (3.7)
NART (Full Scale IQ) [Mean (Standard Deviation); unit: units on a scale] — The National Adult Reading Test (NART) consists of 50 words with irregular phonetic spelling and pronunciation. Score ranges from 0-50, based on the number of words correctly pronounced. The NART score can be used to estimate IQ. Calculating the full scale IQ is done as 127.8-0.78(number of errors on NART). The higher the score, the higher the IQ.
  IQ Scores:
  Over 140 - Genius or near genius. 120 - 140 - Very superior intelligence. 110 - 119 - Superior intelligence. 90 - 109 - Normal or average intelligence. 80 - 89 - Dullness. 70 - 79 - Borderline deficiency.
  units on a scale | 108.0 (9.5) | 102.7 (6.6) | 105.5 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Dementia Rating Scale (DRS) Memory Subscore
Description: The DRS is comprised of: Attention (ATT, 8 items); Initiation-Perseveration (I-P, 11 items); Construction (CONST, 6 items); Conceptualization (CONCEPT, 6 items); and Memory (MEM, 5 items). For this study, only the memory subscore was used, with score possibilities ranging from 0-5, with 5 meaning memory was perfect, 0 being no ability to recall. A negative score indicates a decrease in memory from baseline to 24 weeks.
Time Frame: change from baseline to 24 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Memantine | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
units on a scale | 1.6 [-0.13 to 3.33] | -1.4 [-3.19 to 0.39]

2. Primary Outcome: CIBIC-Plus Score
Description: CIBIC-Plus is based upon clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of informants. It takes into account a subject's overall function in the cognitive, behavioral and functional activity domains. Scoring is based on an interview with the caregiver and examination of the patient by an independent evaluator, without consulting other information such as cognitive test results. It requires the assessor to consider a number of cognitive, functional, and behavioral areas prior to providing an overall "global" assessment of clinical change. 7-point categorical scale that provides a single global rating of change from baseline.A score of 1 indicates marked improvement;and a score of 7, marked worsening.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Memantine | Placebo Oral Tablet
Number analyzed (Participants) | 10 | 10
Participants
  Very Much Improved | 1 | 0
  Much Improved | 5 | 2
  Minimally Improved | 2 | 1
  No Change | 0 | 3
  Minimally Worse | 2 | 2
  Much Worse | 0 | 2
  Very Much Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Active Memantine | Placebo Oral Tablet
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Memantine (N=10) | Placebo Oral Tablet (N=10)
Incident Concentration Difficulties (Nervous system disorders) | 0 (0) | 1 (1) — UKU Incident Symptoms
Incident Fatigue (General disorders) | 2 (2) | 0 (0)
Incident Sleepiness (General disorders) | 2 (2) | 0 (0)
Incident Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Incident Tension (Psychiatric disorders) | 1 (1) | 1 (1)
Increased Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Incident Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Incident Agitation (Psychiatric disorders) | 2 (2) | 1 (1)
Incident Increased Sleep (General disorders) | 3 (3) | 1 (1)
Incident reduced Sleep (General disorders) | 0 (0) | 4 (4)
Incident Increased Dreaming (Nervous system disorders) | 3 (3) | 2 (2)
Incident Dystonia (Nervous system disorders) | 2 (2) | 1 (1)
Incident Rigidity (Nervous system disorders) | 1 (1) | 2 (2)
Incident Hypokinesia (Nervous system disorders) | 1 (1) | 1 (1)
Incident Hyperkinesia (Nervous system disorders) | 1 (1) | 1 (1)
Incident tremor (Nervous system disorders) | 0 (0) | 1 (1)
Incident Akathisia (Nervous system disorders) | 1 (1) | 1 (1)
Incident Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Incident Imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Incident Paresthesias (Nervous system disorders) | 1 (1) | 0 (0)
Incident Headache (Nervous system disorders) | 0 (0) | 1 (1)
Incident Ocular Accommodation disturbances (Nervous system disorders) | 0 (0) | 2 (2)
Incident Increased Salivatino (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incident reduced Salivation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incident Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Incident Micturation Disturbances (Renal and urinary disorders) | 2 (2) | 0 (0)
Incident Polyuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Incident Orthostatic Dizziness (Cardiac disorders) | 1 (1) | 1 (1)
Incident tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Incident Increased Sweating (General disorders) | 1 (1) | 1 (1)
Incident Shivering (General disorders) | 1 (1) | 2 (2)
Incident Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Incident Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Incident Increased Sexual Desire (General disorders) | 1 (1) | 1 (1)
Incident Diminished Sexual Desire (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes